CLINICAL TRIAL: NCT00670748
Title: Phase II Study of Metastatic Cancer That Expresses NY-ESO-1 Using Lymphodepleting Conditioning Followed by Infusion of Anti-NY ESO-1 TCR-Gene Engineered Lymphocytes
Brief Title: Chemotherapy Followed by ESO-1 Lymphocytes and Aldesleukin to Treat Metastatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A more highly selected protocol with ESO TCR opened for pts with melanoma
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 080121; 08-C-0121
Record Dates: First submitted 2008-05-01; First posted 2008-05-02 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Melanoma; Metastatic Renal Cell Cancer; Metastatic Cancer
Keywords: Metastatic Cancer; Gene Therapy; Immunotherapy; Tumor Regression; Metastatic Melanoma; Metastatic Renal Cell Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — aldesleukin; Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- #1 Anti-NY-ESO-1 TCR PBL+HD IL-2 Mel/RCC (Experimental): Patients with melanoma or renal cell cancer (RCC) will receive non-myeloablative lymphodepleting regimen of cyclophosphamide and fludarabine followed by anti-NY ESO-1 T-cell receptor (TCR) peripheral blood lymphocytes (PBL) and high dose aldesleukin.
  Interventions: Biological: Anti-NY ESO-1 T-cell receptor PBL; Drug: aldesleukin; Drug: Cyclophosphamide; Drug: fludarabine phosphate
- #2 Anti-NY-ESO-1 TCR PBL+HD IL-2 OtherCa (Experimental): Patients with cancers other than melanoma or RCC will receive non-myeloablative lymphodepleting regimen of cyclophosphamide and fludarabine followed by anti-NY ESO-1 TCR PBL and high dose (HD) aldesleukin
  Interventions: Biological: Anti-NY ESO-1 T-cell receptor PBL; Drug: aldesleukin; Drug: Cyclophosphamide; Drug: fludarabine phosphate
- #3ESO1 TCR PBL+ALVAC ESO1+HD IL2 Mel/RCC (Experimental): Patients with melanoma or RCC will receive non-myeloablative lymphodepleting regimen of cyclophosphamide and fludarabine followed by replication-defective recombinant canarypox virus (ALVAC) NY-ESO-1 vaccine, anti-NY ESO-1 TCR PBL and high dose aldesleukin
  Interventions: Biological: Anti-NY ESO-1 T-cell receptor PBL; Drug: aldesleukin; Drug: Cyclophosphamide; Drug: fludarabine phosphate; Biological: ALVAC NY ESO-1 vaccine
- #4ESO1 TCR PBL+ALVAC ESO1+HD IL2 OtherCa (Experimental): Patients with cancers other than melanoma or RCC will receive non-myeloablative lymphodepleting regimen of cyclophosphamide and fludarabine followed by ALVAC NY-ESO-1 vaccine, anti-NY ESO-1 TCR PBL and high dose aldesleukin
  Interventions: Biological: Anti-NY ESO-1 T-cell receptor PBL; Drug: aldesleukin; Drug: Cyclophosphamide; Drug: fludarabine phosphate; Biological: ALVAC NY ESO-1 vaccine

INTERVENTIONS:
Biological: Anti-NY ESO-1 T-cell receptor PBL — Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of anti-NY ESO-1 T-cell receptor (TCR) peripheral blood lymphocytes (PBL) and high dose aldesleukin. On day 0,cells (1x10e8 to 1x10e11)will be infused intravenously on the Patient Care Unit over 20-30 minutes.
Drug: aldesleukin — Aldesleukin 720,000 IU/kg intravenous (IV) (based on total body weight)over 15 minutes every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days(maximum of 15 doses)
  Other Names: Proleukin
Drug: Cyclophosphamide — Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml dextrose 5% in water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Other Names: Cytoxan
Drug: fludarabine phosphate — Fludarabine 25 mg/m2/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days.
  Other Names: Fludara
Biological: ALVAC NY ESO-1 vaccine — Approximately two hours prior to cell infusion, patients will receive 0.5 mL containing a target dose of 10e7 cell culture infectious dose 50 (CCID50) (with a range of approximately 10e6.4 to 10e7.9 / mL) of the ESO-1 ALVAC virus S.C. in each extremity (total of 4 x 10e7 CCID50/2 mL.
  Arms: #3ESO1 TCR PBL+ALVAC ESO1+HD IL2 Mel/RCC; #4ESO1 TCR PBL+ALVAC ESO1+HD IL2 OtherCa

SUMMARY:
Background:

-This study uses an experimental cancer treatment that uses the patient s own lymphocytes (type of white blood cell), which are specially selected and genetically modified to target and destroy their tumor.

Objectives:

-To test the safety of the treatment and determine if it can cause the patient s tumor to shrink.

Eligibility:

* Patients greater than 18 years and less than or equal to 66 years of age whose cancer has spread beyond the original site and does not respond to standard treatment.
* Patients have tissue type human leukocyte antigen (HLA)-A*0201.
* Patients cancer cells have the ESO-1 gene.

Design:

* Workup: Patients have scans, x-rays, laboratory tests, and other tests as needed.
* Patients have leukapheresis to collect cells for laboratory treatment and later reinfusion. For this procedure, whole blood is collected thorough a tube in a vein, the desired cells are extracted from the blood, and the rest of the blood is returned to the patient.
* Chemotherapy: Patients have low-dose chemotherapy for 1 week to prepare the immune system to receive the treated lymphocytes.
* Cell infusion and aldesleukin (IL-2) treatment: Patients receive the lymphocytes by a 30-minute infusion through a vein. Starting within 24 hours of the infusion, they receive high-dose aldesleukin infusions every 8 hours for up to 5 days (maximum15 doses).
* Recovery: Patients rest for 1 to 2 weeks to recover from the effects of chemotherapy and aldesleukin.
* Tumor biopsy: Patients may be asked to undergo a biopsy (surgical removal of a small piece of tumor) after treatment to look at the effects of treatment on the immune cells in the tumor.
* Follow-up: After treatment is completed, patients return to the clinic once a month for several months for physical examinations, a review of side effects, laboratory tests and scans. They may undergo leukapheresis at some visits to look at the effect of treatment on the immune system and check the viability of the infused cells. Patients then return to the National Institute of Health (NIH) clinic once a year for 5 years and then complete a follow-up questionnaire for another 10 years.
* Retreatment: Patients whose tumor shrinks or disappears following treatment and then recurs may receive one additional treatment, using the same regimen of chemotherapy, lymphocyte infusion and IL-2 treatment.

DETAILED DESCRIPTION:
Background:

* We have constructed a single retroviral vector that contains both alpha and beta chains of a T cell receptor (TCR) that recognizes the NY-ESO-1 (ESO) tumor antigen, which can be used to mediate genetic transfer of this TCR with high efficiency (> 30%) without the need to perform any selection.
* In co-cultures with human leukocyte antigen serotype within HLA-A A serotype group (HLA-A2) and ESO double positive tumors, anti-ESO TCR transduced T cells secreted significant amount of interferon (IFN)-gamma and additional secretion of cytokines with high specificity.
* Poxviruses encoding tumor antigens, similar to the replication-defective recombinant canarypox virus (ALVAC) ESO-1 vaccine have been shown to successfully immunize patients against these antigens.

Objectives:

Primary objectives:

* Determine if the administration of anti-ESO TCR engineered peripheral blood lymphocytes (PBL) and aldesleukin to patients following a nonmyeloablative but lymphoid depleting preparative regimen will result in clinical tumor regression in patients with metastatic cancer that expresses the ESO antigen.
* Determine if the administration of anti-ESO TCR engineered peripheral blood lymphocytes (PBL), aldesleukin, and ALVAC ESO-1 vaccine to patients following a nonmyeloablative but lymphoid depleting preparative regimen will result in clinical tumor regression in patients with metastatic cancer that expresses the ESO antigen.

Secondary objectives:

* Determine the in vivo survival of TCR gene-engineered cells.
* Determine the toxicity profile of this treatment regimen.

Eligibility:

* Patients who are HLA-A*0201 positive and 18 years of age or older must have:

  * metastatic cancer whose tumors express the ESO antigen;
  * previously received and have been a non-responder to or recurred to standard care for metastatic disease, except for melanoma patients;
* Patients may not have:

  * contraindications for high dose aldesleukin administration.

Design:

* Peripheral blood mononuclear cells (PBMC) obtained by leukapheresis (approximately 5 X 10(9) cells) will be cultured in the presence of anti-cluster of differentiation 3 (CD3) (OKT3) and aldesleukin in order to stimulate T-cell growth.
* Transduction is initiated by exposure of approximately 10(8) to 5 X 10(8) cells to retroviral vector supernatant containing the anti-ESO TCR genes.
* Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of ex vivo tumor reactive, TCR gene transduced PBMC plus intravenous (IV) aldesleukin (720,000 IU/kg q8h for a maximum of 15 doses) with or without ALVAC ESO-1 vaccine. Subcutaneous injection of ALVAC ESO-1 vaccine will be administered on day 0 approximately 2 hours prior to intravenous infusion of cells and a second dose of ALVAC ESO-1 vaccine is given on day 14 (+/- 2 days).
* Patients will undergo complete evaluation of tumor with physical examination, computed tomography (CT) of the chest, abdomen and pelvis and clinical laboratory evaluation four to six weeks after treatment. If the patient has stable disease (SD) or tumor shrinkage, repeat complete evaluations will be performed every 1-3 months. After the first year, patients continuing to respond will continue to be followed with this evaluation every 3-4 months until off study criteria are met.

Cohorts 1 and 2:

* Patients will be entered into two cohorts based on histology: cohort 1 will include patients with metastatic melanoma or renal cell cancer; cohort 2 will include patients with other types of metastatic cancer.
* For each of the 2 strata evaluated, the study will be conducted using a phase II optimal design where initially 21 evaluable patients will be enrolled. For each of these two arms of the trial, if 0 or 1 of the 21 patients experiences a clinical response, then no further patients will be enrolled but if 2 or more of the first 21 evaluable patients enrolled have a clinical response, then accrual will continue until a total of 41 evaluable patients have been enrolled in that stratum.
* For both strata, the objective will be to determine if the combination of high dose aldesleukin, lymphocyte depleting chemotherapy, and anti-ESO TCR-gene engineered lymphocytes is able to be associated with a clinical response rate that can rule out 5% (p0=0.05) in favor of a modest 20% partial response (PR) + complete response (CR) rate (p1=0.20).

Cohorts 3 and 4:

* For patients receiving ALVAC ESO-1 vaccine, patients will also be entered into two cohorts based on histology: cohort 3 for patients with metastatic melanoma or renal cell cancer and cohort 4 for patients with other histologies and all patients will receive the treatment regimen including the ALVAC ESO-1 vaccine.
* For each of these 2 new strata, the study will be conducted using a phase II optimal design where initially 21 evaluable patients will be enrolled. For each of these two new cohorts of the trial, if 0 or 1 of the 21 patients experiences a clinical response, then no further patients will be enrolled but if 2 or more of the first 21 evaluable patients enrolled have a clinical response, then accrual will continue until a total of 41 evaluable patients have been enrolled in that stratum.
* For both strata, the objective will be to determine if the combination of high dose aldesleukin, lymphocyte depleting chemotherapy, anti-ESO TCR-gene engineered lymphocytes, and ALVAC ESO-1 vaccine is able to be associated with a clinical response rate that can rule out 5% (p0=0.05) in favor of a modest 20% PR + CR rate (p1=0.20).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Metastatic cancer that expresses ESO as assessed by one of the following methods: reverse transcription-polymerase chain reaction (RT-PCR) on tumor tissue, or by immunohistochemistry of resected tissue, or serum antibody reactive with ESO. Metastatic cancer diagnosis will be confirmed by the Laboratory of Pathology at the National Cancer Institute (NCI).
* Patients with histologies other than metastatic melanoma, must have previously received systemic standard care (or effective salvage chemotherapy regimens) for metastatic disease, if known to be effective for that disease, and have been either non-responders (progressive disease) or have recurred.
* Greater than or equal to 18 years of age. and less than or equal to 66 years of age.
* Willing to sign a durable power of attorney.
* Able to understand and sign the Informed Consent Document.
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
* Life expectancy of greater than three months.
* Patients of both genders must be willing to practice birth control for four months after receiving the preparative regimen.
* Patients must be human leukocyte antigen (HLA)-A*0201 positive
* Serology:

  * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
  * Seronegative for hepatitis B antigen and hepatitis C antibody unless antigen negative. If hepatitis C antibody test is positive, then patients must be tested for the presence of antigen by RT-PCR and be hepatitis C virus ribonucleic acid (HCV RNA) negative.
* Hematology:

  * Absolute neutrophil count greater than 1000/mm(3) without the support of filgrastim.
  * White blood cell (WBC) (greater than 3000/mm(3)).
  * Platelet count greater than 100,000/mm(3).
  * Hemoglobin greater than 8.0 g/dl.
* Chemistry:

  * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less or equal to 2.5 times the upper limit of normal.
  * Serum creatinine less than or equal to 1.6 mg/dl.
  * Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilberts Syndrome who must have a total bilirubin less than 3.0 mg/dl.
* More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).
* Six weeks must have elapsed since prior ipilimumab therapy to allow antibody levels to decline.
* Patients who have previously received ipilimumab or ticilimumab anti-programmed cell death protein 1 (PD1) or anti-PD-L1 antibodies, and have documented gastrointestinal (GI) toxicity must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

* Prior vaccination with an replication-defective recombinant canarypox virus (ALVAC) containing vaccine for patients who will receive the ALVAC ESO-1 vaccine (cohorts 3 or 4).
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
* Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* Concurrent Systemic steroid therapy.
* Known systemic hypersensitivity to any of the vaccine components, including egg products or Neomycin for patients who will receive the ALVAC ESO-1 vaccine (cohorts 3 or 4).
* History of severe immediate hypersensitivity reaction to any of the agents used in this study.
* History of coronary revascularization or ischemic symptoms.
* Any patient known to have an left ventricular ejection fraction (LVEF) less than or equal to 45 percent.
* Documented forced expiratory volume (LVEF) of less than or equal to 45 percent tested in patients with:

  * History of ischemic heart disease, chest pain, or clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block.
  * Age greater than or equal to 60 years old.
* Documented forced expiratory volume in 1 second (FEV1) less than or equal to 60 percent predicted tested in patients with:

  * A prolonged history of cigarette smoking (20 pk/year of smoking within the past 2 years).
  * Symptoms of respiratory dysfunction

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-05-29 (Actual); Primary Completion 2016-06-29 (Actual); Study Completion 2016-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeng G, Touloukian CE, Wang X, Restifo NP, Rosenberg SA, Wang RF. Identification of CD4+ T cell epitopes from NY-ESO-1 presented by HLA-DR molecules. J Immunol. 2000 Jul 15;165(2):1153-9. doi: 10.4049/jimmunol.165.2.1153. PMID 10878395
- [Background] Zhao Y, Bennett AD, Zheng Z, Wang QJ, Robbins PF, Yu LY, Li Y, Molloy PE, Dunn SM, Jakobsen BK, Rosenberg SA, Morgan RA. High-affinity TCRs generated by phage display provide CD4+ T cells with the ability to recognize and kill tumor cell lines. J Immunol. 2007 Nov 1;179(9):5845-54. doi: 10.4049/jimmunol.179.9.5845. PMID 17947658
- [Background] Valmori D, Dutoit V, Lienard D, Rimoldi D, Pittet MJ, Champagne P, Ellefsen K, Sahin U, Speiser D, Lejeune F, Cerottini JC, Romero P. Naturally occurring human lymphocyte antigen-A2 restricted CD8+ T-cell response to the cancer testis antigen NY-ESO-1 in melanoma patients. Cancer Res. 2000 Aug 15;60(16):4499-506. PMID 10969798
- [Derived] Crompton JG, Sukumar M, Roychoudhuri R, Clever D, Gros A, Eil RL, Tran E, Hanada K, Yu Z, Palmer DC, Kerkar SP, Michalek RD, Upham T, Leonardi A, Acquavella N, Wang E, Marincola FM, Gattinoni L, Muranski P, Sundrud MS, Klebanoff CA, Rosenberg SA, Fearon DT, Restifo NP. Akt inhibition enhances expansion of potent tumor-specific lymphocytes with memory cell characteristics. Cancer Res. 2015 Jan 15;75(2):296-305. doi: 10.1158/0008-5472.CAN-14-2277. Epub 2014 Nov 28. PMID 25432172
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-C-0121.html

RESULTS

PARTICIPANT FLOW:
Groups:
- #1 Anti-NY-ESO-1 TCR PBL+HD IL-2 Mel/RCC; #2 Anti-NY-ESO-1 TCR PBL+HD IL-2 OtherCa: Biological/Vaccine: Anti-NY ESO-1 T-cell receptor PBL Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of anti-NY ESO-1 T-cell receptor (TCR) peripheral blood lymphocytes (PBL) and high dose aldesleukin. On day 0,cells (1x10e8 to 1x10e11)will be infused intravenously on the Patient Care Unit over 20-30 minutes.
  Drug: aldesleukin Aldesleukin 720,000 IU/kg intravenous (IV) (based on total body weight)over 15 minutes every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days(maximum of 15 doses) Drug: Cyclophosphamide Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml dextrose 5% in water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Drug: fludarabine phosphate Fludarabine 25 mg/m2/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days.
- #3ESO1 TCR PBL+ALVAC ESO1+HD IL2 Mel/RCC: Pts will receive non-myeloablative lymphodepleting prep regimen:cyclophosphamide & fludarabine followed by the anti-NY ESO-1 T-cell receptor (TCR) peripheral blood lymphocytes (PBL) & high dose aldesleukin. On day 0,cells (1x10e8 to 1x10e11)will be infused intravenously on the Pt Care Unit over 20-30 min. Aldesleukin 720,000 IU/kg intravenous (IV) (based on total body wt)over 15 min. every 8 hrs (+/-1 hr) beginning within 24 hrs of cell infusion and continuing for up to 5 days(max. of 15 doses).Cyclophosphamide 60 mg/kg/dayX2 days IV in 250 ml dextrose 5% in water (D5W) with Mesna 15 mg/kg/dayX2 days over 1 hr.
  Fludarabine 25 mg/m2/day intravenous piggyback (IVPB) daily over 30 min. for 5 days.
  ALVAC NY ESO-1 vaccine:Approx. 2hrs prior to cell infusion, pts will receive 0.5 mL containing a target dose of 10e7 cell culture infectious dose 50 (CCID50)(with a range of approx. 10e6.4 to 10e7.9 / mL) of the ESO-1 ALVAC virus S.C. in each extremity (total of 4 x 10e7 CCID50/2 mL.
- #4ESO1 TCR PBL+ALVAC ESO1+HD IL2 OtherCa: Anti-NY ESO-1 T-cell receptor PBL; Pts will receive non-myeloablative lymphodepleting prep regimen cyclophosphamide and fludarabine followed by anti-NY ESO-1 T-cell receptor (TCR) peripheral blood lymphocytes (PBL) and high dose aldesleukin. On day 0,cells (1x10e8 to 1x10e11)will be infused intravenously on the Pt Care Unit over 20-30 min. Aldesleukin 720,000 IU/kg IV (based on total body wt)over 15 min. every 8 hours (+/-1 hr) beginning within 24 hrs of cell infusion and continuing for up to 5 days(max. of 15 doses). Cyclophosphamide 60 mg/kg/dayX2 days IV in 250 ml dextrose 5% in water (D5W) with Mesna 15 mg/kg/dayX2 days over 1 hr. Fludarabine 25 mg/m2/day IVPB daily over 30 min. for 5 days. ALVAC NY ESO-1 vaccine:Approx. 2 hrs prior to cell infusion, patients will receive 0.5 mL containing a target dose of 10e7 cell culture infectious dose 50 (CCID50) (with a range of approx.10e6.4 to 10e7.9 / mL) of the ESO-1 ALVAC virus S.C. in each extremity (total of 4 x 10e7 CCID50/2 mL.
Period: Overall Study
Arm/Group | #1 Anti-NY-ESO-1 TCR PBL+HD IL-2 Mel/RCC | #2 Anti-NY-ESO-1 TCR PBL+HD IL-2 OtherCa | #3ESO1 TCR PBL+ALVAC ESO1+HD IL2 Mel/RCC | #4ESO1 TCR PBL+ALVAC ESO1+HD IL2 OtherCa
Started | 17 | 16 | 7 | 5
Completed | 14 | 14 | 5 | 4
Not Completed | 3 | 2 | 2 | 1
Not completed — Death during treatment | 1 | 1 | 1 | 0
Not completed — Not off study | 2 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | #1 Anti-NY-ESO-1 TCR PBL+HD IL-2 Mel/RCC | #2 Anti-NY-ESO-1 TCR PBL+HD IL-2 OtherCa | #3ESO1 TCR PBL+ALVAC ESO1+HD IL2 Mel/RCC | #4ESO1 TCR PBL+ALVAC ESO1+HD IL2 OtherCa | Total
Number analyzed (Participants) | 17 | 16 | 7 | 5 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 7 | 5 | 42
  >=65 years | 1 | 2 | 0 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (11.6) | 38.9 (14.1) | 44.4 (10.4) | 38.8 (16.0) | 43.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 2 | 2 | 16
  Male | 12 | 9 | 5 | 3 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 0 | 4
  Not Hispanic or Latino | 15 | 15 | 6 | 5 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 15 | 14 | 6 | 5 | 40
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 16 | 7 | 5 | 45

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Per the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Response was determined by the RECIST. Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Progressive disease (PD) is at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD.
Time Frame: Approximately 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | #1 Anti-NY-ESO-1 TCR PBL+HD IL-2 Mel/RCC | #2 Anti-NY-ESO-1 TCR PBL+HD IL-2 OtherCa | #3ESO1 TCR PBL+ALVAC ESO1+HD IL2 Mel/RCC | #4ESO1 TCR PBL+ALVAC ESO1+HD IL2 OtherCa
Number analyzed (Participants) | 17 | 16 | 7 | 5
Participants
  Complete Response | 3 | 1 | 1 | 0
  Partial Response | 6 | 7 | 1 | 3
  Progressive Disease | 7 | 7 | 4 | 2
  Stable Disease | 0 | 0 | 0 | 0
  Not Evaluable | 1 | 1 | 1 | 0

2. Secondary Outcome: Number of Participants With In Vivo Survival of T-Cell Receptor (TCR)-Engineered Cells
Description: Immunological monitoring using both tetramer analysis and staining for the T cell receptor (TCR). This will provide data to estimate the in vivo survival of lymphocytes derived from the infused cells.
Time Frame: 1 month post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | #1 Anti-NY-ESO-1 TCR PBL+HD IL-2 Mel/RCC | #2 Anti-NY-ESO-1 TCR PBL+HD IL-2 OtherCa | #3ESO1 TCR PBL+ALVAC ESO1+HD IL2 Mel/RCC | #4ESO1 TCR PBL+ALVAC ESO1+HD IL2 OtherCa
Number analyzed (Participants) | 17 | 16 | 7 | 5
Participants | 16 | 16 | 6 | 4

3. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately, 66 months and 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | #1 Anti-NY-ESO-1 TCR PBL+HD IL-2 Mel/RCC | #2 Anti-NY-ESO-1 TCR PBL+HD IL-2 OtherCa | #3ESO1 TCR PBL+ALVAC ESO1+HD IL2 Mel/RCC | #4ESO1 TCR PBL+ALVAC ESO1+HD IL2 OtherCa
Number analyzed (Participants) | 17 | 16 | 7 | 5
Participants | 17 | 16 | 7 | 5

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately, 66 months and 10 days.
Arm/Group | #1 Anti-NY-ESO-1 TCR PBL+HD IL-2 Mel/RCC | #2 Anti-NY-ESO-1 TCR PBL+HD IL-2 OtherCa | #3ESO1 TCR PBL+ALVAC ESO1+HD IL2 Mel/RCC | #4ESO1 TCR PBL+ALVAC ESO1+HD IL2 OtherCa
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16 | 1/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/17 | 3/16 | 2/7 | 2/5
Other Adverse Events (participants affected / at risk) | 17/17 | 16/16 | 7/7 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | #1 Anti-NY-ESO-1 TCR PBL+HD IL-2 Mel/RCC (N=17) | #2 Anti-NY-ESO-1 TCR PBL+HD IL-2 OtherCa (N=16) | #3ESO1 TCR PBL+ALVAC ESO1+HD IL2 Mel/RCC (N=7) | #4ESO1 TCR PBL+ALVAC ESO1+HD IL2 OtherCa (N=5)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Death not associated with CTCAE term (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | #1 Anti-NY-ESO-1 TCR PBL+HD IL-2 Mel/RCC (N=17) | #2 Anti-NY-ESO-1 TCR PBL+HD IL-2 OtherCa (N=16) | #3ESO1 TCR PBL+ALVAC ESO1+HD IL2 Mel/RCC (N=7) | #4ESO1 TCR PBL+ALVAC ESO1+HD IL2 OtherCa (N=5)
Hemoglobin (Blood and lymphatic system disorders) | 15 (15) | 14 (14) | 4 (4) | 4 (4)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 17 (17) | 16 (16) | 7 (7) | 5 (5)
Lymphopenia (Blood and lymphatic system disorders) | 17 (17) | 16 (16) | 7 (7) | 5 (5)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 17 (17) | 16 (16) | 7 (7) | 5 (5)
Platelets (Blood and lymphatic system disorders) | 14 (14) | 16 (16) | 6 (6) | 5 (5)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0x10e9/L) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, GI (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hemorrhage/Bleeding - Other (Hemorrhage sub-retinal OS) (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Infections and infestations) | 12 (12) | 13 (13) | 5 (5) | 4 (4) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0x10e9/L, fever >/=38.5 degrees C)
Infection (Infections and infestations) | 5 (5) | 4 (4) | 1 (1) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5 (5) | 6 (6) | 1 (1) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 1 (1) | 2 (2)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 5 (5) | 11 (11) | 4 (4) | 2 (2)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal/Soft Tissue - Other (fracture: right acetabulum) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Pain (General disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 10 (10) | 3 (3) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8) | 2 (2) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal/Genitourinary - Other (low urine output) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute vascular leak syndrome (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
PTT (Partial Thromoboplastin Time) (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CD4 count (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-07-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT00670748/Prot_SAP_000.pdf
  • Informed Consent Form (2015-07-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT00670748/ICF_001.pdf